#### VA RESEARCH CONSENT FORM

| Subject Name: | | Date: _ | |
|---|---|---|---|
| Title of Study: Compre | hensive Wide Bandwidth Test B | attery of Auditory Function in Vete | erans |
| Principal Investigator: | Kim S. Schairer, Ph.D. | VAMC: James H. Quil | len VAMC |
| This Informed Consent will ex you read this material carefully | | | important that |
| PURPOSE | | | |
| The purpose of this research prinvestigational device that test the currently-used clinical equacross a wider range of sound determine whether the current hearing loss and middle ear dy | s inner ear, middle ear, and a ipment. This new device will a lis than the range used with call and new devices are the sar | auditory brainstem function wit<br>allow us to measure how soun<br>urrent clinical equipment. Our | h results from<br>d is transmitted<br>goal is to |
| DURATION | | | |
| The expected duration of study | y participation is up to three h | ours. | |
| PROCEDURES | | | |
| The procedures which will invo | olve you as a research subjec | et include: | |
| Chart Review: If you agree to your ear health (e.g., from pring gathered from your medical reenrolled at the Mountain Home included in the study. | nary care, emergency room, on<br>cord. If your medical record is | or ear, nose, and throat doctor<br>s not available (i.e., you are no | s) will be<br>It a Veteran |
| | | ā. | |
| UBJECT'S IDENTIFICATION (I.D. plate of g | give name - last, first, middle) | | |
| | | Subject's Initials | |
| | | VA FORM | |

James H. Quillen VAMC

Version Date: 01/16/2019
Approved by ETSU/VA Medical IRB / Approval Date: October 17,
DSC 151-115-004
2019 / Expiration Date: October 16, 2020
April 1991 (RS) 10-1086

#### VA RESEARCH CONSENT FORM

(Continuation )

| Subject Name: | | Date: |
|---|---|---|
| Title of Study: Comprehe | ensive Wide Bandwidth Test | t Battery of Auditory Function in Veterans |
| Principal Investigator:_ | Kim S. Schairer, Ph.D. | VAMC: James H. Quillen VAMC |
| Clinical procedure. Otoscopy of There are no known risks for to tooscope tip) in your ear can to have them cleaned before an ear, nose, and throat doctors. | will take approximately two this procedure, except poo al. If your ear canals are to participating in the study. or if there is evidence of d may be asked to return a | canals using an otoscope. This is a standard or minutes, and all you have to do is sit quietly. ssible discomfort with placement of the speculum blocked with cerumen (earwax), you may be asked You will be referred to your primary care doctor or trainage or another sign that may be associated and continue your participation after you see the |
| performed in the Audiology cli<br>ears and respond 'yes' when<br>There are no known risks for<br>hearing test results unless you<br>you have a hearing loss, and | inic. You will be asked to a<br>you hear soft tones. The t<br>taking this test. You will no<br>u were specifically recruite<br>we do not currently need | pure tone hearing threshold test, like those sit in a quiet room with insert earphones in your test will take approximately 20 to 30 minutes. To be excluded from the study based on your ed for a normal hearing group, the results indicate subjects in the groups with hearing loss. If a new you will be referred to an audiologist. |
| you will be asked to repeat we which volume the words become they will be in the same local | ords at soft levels, repeat<br>me uncomfortably loud. T<br>ion and use the same equ | clinical speech audiometry tests. For these tests, words at a comfortable volume, and indicate at These tests will take approximately 15 minutes. uipment as the pure tone hearing test. There are xcluded from the study based on these test |
| tests give us information about (acoustic reflex threshold test approximately 10 minutes. Duplastic probe tip in each ear, for you do not like the feeling of properties. | ut well your middle ears (to<br>) are working. This set of<br>uring the tests, all you will<br>feel some pressure in you<br>pressure in your ear canal | receive a standard clinical test battery. These sympanometry test) and middle ear muscles tests will be completed in a quiet room and take be asked to do is sit quietly. You will have a small ar ear canals, and hear several different beeps. If its or feel uncomfortable during this test, please tell not be excluded from the study based on the |
| V | | |
| Version Date: 01/16/2019 | | Subject's Initials |

#### VA RESEARCH CONSENT FORM

(Continuation )

| Subject Name: | Date: |
|---|---|
| Title of Study: Comprehensive Wide Bandwidth Test Battery | of Auditory Function in Veterans |
| Principal Investigator: Kim S. Schairer, Ph.D. | VAMC: James H. Quillen VAMC |
| Experimental Immittance Test Battery: This test is similar to battery, but it is completed using experimental equipment and environment, expectations for you, and risks are the same as t not be excluded from the study based on the results of this test. Otoacoustic Emissions (OAE): You will receive an OAE test. | the sounds will be different. The test hose stated for the Standard test. You will t. |
| as the Experimental immittance test battery. The OAE test tells You will be asked to sit quietly for approximately 10 minutes will completed in a quiet room, and you will hear some sounds through the are no known risks from taking this test. You will not be test results. | s us how well your inner ears are working.<br>hile the test is completed. The test will be<br>ough a foam probe tip in your ear canal. |
| ALTERNATIVE PROCEDURES/TREATMENTS | |
| The alternative procedures/treatments available to you if you e alternative to the experimental test is the clinical test, which is as a typical hearing test in the Audiology clinic. | lect not to participate in this study are: The part of both this research protocol as well |
| POSSIBLE RISKS/DISCOMFORTS | |
| The possible risks and/or discomforts of your involvement included otoscope speculum, discomfort from the probes used for the clear tests, discomfort with pressure in the ear canals during the sounds used in the middle ear and speech tests. If you are undof the tests, please tell the researcher and he or she will stop the expected risks from the tests included in this study. | inical and experimental middle and inner se tests, and loudness discomfort from the comfortable and/or want to stop during any |
| Version Date: 01/16/2019 | Subject's Initials |

#### VA RESEARCH CONSENT FORM

(Continuation )

| Subject Name: Title of Study: Comprehensive Wide Bandwidth Test Battery of Auditory Function in Veterans Principal Investigator: Kim S. Schairer, Ph.D. VAMC: James H. Quillen VAMC |
|---|
| POSSIBLE BENEFITS The possible benefits of your participation are: Benefits to you include the knowledge that you are making valuable contributions toward the application of new tests of inner ear and middle ear function in clinical practice. If a previously unidentified hearing loss is found, you will receive counseling and an audiologist and/or an ear, nose, and throat doctor will be recommended. If you have a previously diagnosed hearing loss, your participation in the study may provide you with additional information about |
| your hearing. The proposed research may lead to better measurement procedures and clinical devices that could be used to improve the quality of screening and diagnostic procedures to detect inner and middle ear problems and related hearing loss in Veterans. INJURY/COMPLICATIONS |
| For studies being conducted at the James H. Quillen VA Medical Center: |
| According to VA Regulations [38CFR17.85 (a)] the medical facility shall provide necessary medical treatment to a research subject injured as a result of participation in a research project (unless the injury is a result of not following study procedures). However, no additional compensation has been set aside. You have not waived any legal rights or released the VA or its agents from liability for negligence by signing this form. |
| FINANCIAL COSTS |
| Some veterans are required to pay copayments for medical care and services provided by VA. These copayment requirements will continue to apply to medical care and service provided by VA that are not part of this study. |
| There are no financial costs to you for participating in this study. |
| COMPENSATION IN THE FORM OF PAYMENTS TO RESEARCH SUBJECTS |
| You will be compensated \$25 for your involvement in this study. |
| Version Date: 01/16/2019 Subject's Initials |

#### VA RESEARCH CONSENT FORM

(Continuation )

| Subject Name: Title of Study: Comprehensive Wide Bandwidth Test Battery of Auditory Function in Veterans |
|---|
| Principal Investigator: Kim S. Schairer, Ph.D. VAMC: James H. Quillen VAMC |
| VAMC: James H. Quillen VAMC VAMC: James H. Quillen VAMC VAMC: James H. Quillen VAMC VAMC: James H. Quillen VAMC VAMC: James H. Quillen VAMC Participation in this research experiment is voluntary. You may refuse to participate and may quit at any time. If you quit or refuse to participate, the benefits or treatment to which you are entitled will not be affected. You may quit during any of the tests, or by calling Dr. Kim Schairer at 423-926-1171 ext. 7138. If any of the research results may lead you to change your mind about staying in the study, you will be informed right away. The Principal Investigator may take you out of the study at any time without your consent if he or she decides that it is not in your best interest to continue (i.e., not following study-related directions, adverse event). You may also be taken off the study if it ends early. If there may be any adverse consequences (physical/social/economic, legal, or psychological), of a participant's decision to withdraw from the research, the consent process must disclose the consequences and procedures for orderly termination of participation. If there are significant new findings are likely during the course of the research which may impact the subject's willingness to continue his or her participation, the consent process must disclose that these new findings will be provided to them. CONTACT FOR QUESTIONS If you have any questions, problems, research-related medical problems, or if you would like to verify the validity of a study, you may contact Dr. Kim S. Schairer at 423-926-1171 ext. 7138 or Mrs. Jeanne Lilly at 423-926-1171 ext. 7555. You may also contact the Chairman of the Institutional Review Board (IRB) at 423-439-6054 for any questions you have about your rights as a research subject. If you have any questions or concerns about the research and want to talk to someone independent of the research team, or if you are unable to reach the study staff, you may call an IRB Coordinator at 423-439-6055 or |
| Version Date: 01/16/2019 Subject's Initials |

#### VA RESEARCH CONSENT FORM

(Continuation )

| Title of Study. | • | ensive Wide Bandwidth Te | est Battery of Auditory | Date: |
|---|---|---|---|---|
| Principal Investig | ator:_ | Kim S. Schairer, Ph.D. | VAMC: | James H. Quillen VAMC |
| from this experiment of accordance with the represented at meetings identifying you as a sustate University (ETS (ORO), General Accordance Research Protection ( | will be steecord cos, share ubject. Tuj/VA If untabilit | tored in the Applied Head<br>ontrol schedule. The resid with clinicaltrials.gov,<br>The study records are ac<br>RB, VA Research & Dev<br>y Office (GAO), Food & | aring Science Lab in sults of this study may and with data collect cessible to the study elopment Committed Drug Administration kept completely co | tion software developers without by personnel, East Tennessee ee, Office of Research Oversight (FDA), and Office of Human offidential according to current |
| Our collaborators, Do Ph.D. at the Portland hearing test data from University (OHSU). The security number, date the date on which you | ug Keef<br>VA Med<br>a a prote<br>nese da<br>of birth<br>a are see | e, Ph.D. at Boys Town I<br>lical Center, as well as t<br>ected computer network<br>ta will not contain perso | National Research Heir study staff, will drive located at Ore nally identifiable informane number). How te on the experimen | Hospital and M. Patrick Feeney, receive your experimental egon Health & Science ormation (e.g., full name, social wever, these data will contain tal system has been |
| data to a network driv<br>Boys Town National F<br>study staff will be resp<br>original research reco<br>accordance with curre<br>at Boys Town National | e at OH<br>Research<br>consible<br>rds, bot<br>ent record<br>al Resea<br>y staff, i | SU. The James H. Quill<br>h Hospital, and M. Patri<br>for maintaining the sec<br>h paper and electronic,<br>rds retention requirement<br>arch Hospital and M. Pa | len VAMC study per<br>ck Feeney, Ph.D. at<br>urity and confidentia<br>will be maintained a<br>nts. Any information<br>trick Feeney, Ph.D. | by of your de-identified research resonnel, Doug Keefe, Ph.D. at the Portland VAMC and their ality of this transferred data. All at the James H. Quillen VAMC in shared with Doug Keefe, Ph.D. at the Portland VA Medical aw. However, this information will |
| Quillen VA Medical C | enter, a | | d dated Consent Fo | in a study at the James H.<br>rm will be placed in your medical<br>our medical record. |
| Version Date: 01/16/2 | 2019 | | | Subject's Initials |

#### VA RESEARCH CONSENT FORM

(Continuation )

| Subject Name: | Date: |
|---|---|
| Title of Study: Comprehensive Wide Bandwidth | Test Battery of Auditory Function in Veterans |
| Principal Investigator: Kim S. Schairer, Ph.D. | VAMC: James H. Quillen VAMC |
| | http://www.ClinicalTrials.gov, as required by United f the results, but will not include information that may ne. |
| CONSENT | |
| | had this document read to me and I have been giver<br>sk questions and to discuss my participation with the<br>I freely and voluntarily choose to participate in this |
| Signature of Subject | Date Last 4 of SSN (MONTH/DAY/YEAR) |
| Signature of Person Obtaining Consent | Date<br>(MONTH / DAY / YEAR) |
| Version Date: 01/16/2019 | Subject's Initials |

| 8 |
|---|

| Subject Name: | Date: |
|---|---|
| Study Title: Comprehensive Wide Bandwidth Test Battery of Aud | itory Function in Veterans |
| VAMC: James H. Quillen VAMC | |

# AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION FOR RESEARCH PURPOSES

The privacy law, Health Insurance Portability & Accountability Act (HIPAA), protects my individually identifiable health information (protected health information). The privacy law requires me to sign an authorization (or agreement) in order for researchers to be able to use or disclose my protected health information for research purposes in the study entitled *Comprehensive Wide Bandwidth Test Battery of Auditory Function in Veterans*.

I authorize Kim S. Schairer, Ph.D. and her research staff to use and disclose my protected health information for the purposes described below. I also permit the research staff to disclose my protected health information for the purposes described below. My protected health information that may be used and disclosed includes:

| √ Names |
|---|
| √ All geographic subdivisions smaller than a state, except for the initial three digits |
| of the zip code if the geographic unit formed by combining all zip codes with the |
| same three initial digits contains more than 20,000 people |
| √ All elements of dates except year for dates directly related to an individual, |
| including birth date, admission date, discharge date, date of death; and all ages over |
| 89 and all elements of dates (including year) indicative of such age, except that such |
| ages and elements may be aggregated into a single category of age 90 or older. |
| √ Telephone numbers |
| ☐ Fax numbers |
| √ E-mail addresses |
| √ Social security numbers |
| √ Medical record numbers |
| ☐ Health plan beneficiary numbers |
| ☐ Account numbers |
| ☐ Certificate or license numbers |
| ☐ Vehicle identifiers and license plate numbers |
| ☐ Device identifiers and serial numbers |
| □ URLs |
| ☐ Internet Protocol (IP) addresses |
| ☐ Biometric identifiers including fingerprints and voiceprints |
| ☐ Full-face photographs and any comparable images |
| ☐ Any other unique, identifying characteristic or code, except as permitted for re- |
| identification in the Privacy Rule |

Health Information that will be collected from the following sources (please check all that apply):

| Sub | ect's | Initial | S |
|-----|-------|-----------|----|
| Duo | CCL 3 | TITICICAL | ., |

Version Date: 10/19/2018

| Subject Name: Date: |
|---|
| Study Title: Comprehensive Wide Bandwidth Test Battery of Auditory Function in Veterans VAMC: James H. Quillen VAMC |
| VANIC: James H. Quillen VANIC |
| √ Review of the electronic Medical Record (CPRS): |
| √ History and Physical Exam: |
| √ Consultation Reports: √ X-ray Reports: |
| ☐ Laboratory tests: |
| √ Operative tests: |
| √ Discharge Summary: |
| √ Progress Notes: |
| √ Questionnaires, interview results, focus group survey, psychology survey, psychological performance tests: |
| Photographs, videotapes, audiotapes, or digital or other images: |
| ☐ Tissue and/or blood specimens: √ Other: |
| v Other. |
| In accordance with 38 USC 7332 (Applicable to Drug Abuse, Alcohol Abuse, HIV Infection, and Sickle Cell Anemia Records). The PI provides assurance in writing that the purpose of the data is to conduct scientific research and that no personnel involved in the study may identify, directly or indirectly, any individual patient or subject in any report of such research or otherwise disclose patient or subject identities in any manner. Please check all that apply: |
| ☐ Acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV) infection. |
| Treatment for drug or alcohol abuse. |
| ☐ Sickle cell anemia. |
| The Investigator, Kim S. Schairer, Ph.D. may use and share my health information with: |
| <ul> <li>The East Tennessee State University Human Research Protections Program (HRPP) Institutional Review Board Administration when the researcher or the research site is undergoing Quality Improvement Program (QIP) auditing.</li> <li>The James H. Quillen Veterans Affairs Medical Center Office of Research &amp; Development when the researcher or the research site is undergoing Quality Improvement Program (QIP) auditing.</li> <li>Government representatives, when required by law</li> <li>Hospital (VAMC or Mountain States Health Alliance) representatives</li> </ul> |
| Once my health information has been disclosed to anyone outside of this study, the information may no longer be protected under this authorization. |
| The investigator(s) Kim S. Schairer, Ph.D. (researcher) agree to protect my health information by using and disclosing it only as permitted by me in this Authorization and as directed by state and federal law. I do not have to sign this Authorization. If I decide not to sign the Authorization: |
| <ul> <li>It will not affect my treatment, payment or enrollment in any health plans nor affect my eligibility<br/>for benefits.</li> </ul> |

Subject's Initials

Version Date: 10/19/2018

| Subject Name:Study Title: Comprehensive Wide Band | width Toet Battory of Au | Date: |
|---|---|---|
| VAMC: James H. Quillen VAMC | width rest battery of Ad | ditory Function in Veterans |
| <ul> <li>I may not be allowed to participate in</li> </ul> | this research study | |
| After signing the Authorization, I can char | nge my mind and: | |
| <ul> <li>Not let the researcher disclose or use my protected health information (revoke the Authorization If I revoke the Authorization, I will send a written letter to: Kim S. Schairer, Audiology (126), James H. Quillen VAMC, P.O. Box 4000, Mountain Home, TN 37684 to inform him/her of my decision.</li> </ul> | | |
| <ul> <li>If I revoke this Authorization, researc<br/>information already collected for this</li> </ul> | | sclose the protected health |
| <ul> <li>If I revoke this Authorization my protestshould I have an adverse event (a base)</li> <li>If I change my mind and withdraw the participate in the study.</li> </ul> | ected health information mad effect, or experience so | mething unanticipated). |
| This Authorization does not have an expiration | on date. | |
| If I have not already received a copy of the<br>Privacy Officer. If I have any questions or<br>VAMC Privacy Officer, Ms. Angela Mullins<br>Tennessee State University, James H. Qui<br>Wright, at (423) 433-6074. | concerns about my priv- Allen, at (423) 926-117 | vacy rights, I should contact the 1, Ext 7620, or the East |
| I am the subject or am authorized to act or<br>I will receive a copy of this form after it is | | I have read this information, and |
| 8 | | |
| | , | |
| Signature of research subject or | Date | Last 4 of SSN |
| Printed name of research subject | | |

Subject's Initials

Version Date: 10/19/2018

| | 8 |
|----|---|
| ŭ. | |
| • | |